CLINICAL TRIAL: NCT05515120
Title: Rivaroxaban Plus Aspirin Versus Acenocoumarol to Manage Recurrent Venous Thromboembolic Events Despite Systemic Anticoagulation With Rivaroxaban
Brief Title: Rivaroxaban Plus Aspirin to Manage Recurrent Venous Thromboembolic Events
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Maximiliano Victor Manuel Correa Lara, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000001
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Venous Thromboembolism; Anticoagulant-induced Bleeding; Venous Thromboses; Pulmonary Embolism
Keywords: venous thromboembolism; Rivaroxaban; Aspirin; Acenocoumarol
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Rivaroxaban; Aspirin; Acenocoumarol; acarboxyprothrombin

STUDY DESIGN:
Intervention Model Description: It was adopted an equal allocation of patients to each treatment (i.e., 1:1 randomization)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rivaroxaban plus Aspirin (Active Comparator): Drug: Rivaroxaban 15 mg Rivaroxaban 15 mg BID
  Other Names:
  Xarelto 15 mg Rivaroxabana 15 mg Drug: Aspirin 300 mg
  Interventions: Drug: Rivaroxaban 20 MG [Xarelto]; Drug: Aspirin 300mg
- Acenocoumarol (Placebo Comparator): Drug: Acenocoumarol Other Name: Vitamin K antagonist
  Interventions: Drug: Acenocoumarol Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 20 MG [Xarelto] — It was adopted an equal allocation of patients to each treatment (i.e., 1:1 randomization)
  Other Names: Xarelto 20 mg
  Arms: Rivaroxaban plus Aspirin
Drug: Aspirin 300mg — It was adopted an equal allocation of patients to each treatment (i.e., 1:1 randomization)
  Other Names: Acetilsalicilic acid
  Arms: Rivaroxaban plus Aspirin
Drug: Acenocoumarol Oral Tablet — It was adopted an equal allocation of patients to each treatment (i.e., 1:1 randomization)
  Other Names: Vitamin K antagonist
  Arms: Acenocoumarol

SUMMARY:
Venous thromboembolism affects around 10 million people per year worldwide, however, despite its high incidence, there is no systematic review or randomized trial focused on the treatment of patients with recurrent deep vein thrombosis (DVT) and/or or pulmonary embolism (PE) during anticoagulant treatment. The objective was to compare the use of Rivaroxaban plus Aspirin versus Acenocoumarol in patients with recurrent venous thromboembolism treated with rivaroxaban.

DETAILED DESCRIPTION:
Venous thromboembolism has two manifestations, deep vein thrombosis (DVT) and pulmonary embolism (PE), affects around 10 million people per year worldwide, with an annual incidence of 1-2 cases per 1000 population and increases exponentially with age. [1,2,3] DVT is a multicausal disease thought to be triggered by interactions between multiple triggering factors that may be additive or synergistic, such as active cancer, antiphospholipid syndrome (APS), or other chronic inflammatory disorders. [2,4] The contribution of genetics to the risk of thromboembolism venous traditionally includes protein C, protein S, and antithrombin deficiencies, prothrombin gene mutation, and factor V Leiden. [5] The exact epidemiology in Mexico is unknown, however, the estimated prevalence of deficiencies in a population studied in Mexico City were Protein C (PC) 0.65%, Protein S (PS) 0.65%, Antithrombin (AT) 2.04% and Plasminogen ( Plg) 2.5%. [6] For the treatment of patients with DVT and/or PE, the American Society of Hematology (ASH) guideline panel suggests using direct oral anticuagulants (DOACs) over vitamin K antagonists (VKAs), [7] however the use of a DOAC instead of a VKA for patients with DVT does not impact mortality, the use of DOACs has also been related to a reduction in the risk of DVT and major bleeding, although this was not statistically significant, the greatest advantage is that the use of DOACs do not require frequent dose adjustment, monitoring of the INR, or dietary restrictions, [8 -31] in our work center we started with DOACs as the first line of treatment.

Recurrent DVT despite anticoagulation has been related to the presence of active cancer, subtherapeutic anticoagulation, use of concomitant anticancer drugs, younger age at presentation (<65 years), and PE as the initial DVT. [32-40] Insertion of an inferior vena cava (IVC) filter was previously recommended in patients with recurrent DVT while receiving anticoagulant therapy. [41] However, the risk of recurrent DVT after IVC filter insertion is as high as 32% in cancer patients and has been associated with significant morbidity and poor quality of life; [42-46] It has been suggested that increasing the dose of low molecular weight heparin (LMWH) may be an alternative to IVC filter insertion in patients with recurrent DVT, [47-49] however, to date, there is no systematic review or randomized trial focused on the treatment of patients with recurrent DVT and/or PE during anticoagulant treatment.

The aim of the current study was to compare the use of Rivaroxaban plus Aspirin versus Acenocoumarol in the prevention of thromboembolic and bleeding events in patients with recurrent venous thromboembolism treated with rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

Objectively proven first episode of venous thromboembolism (upper extremity deep vein thrombosis, proximal lower extremity deep vein thrombosis, or pulmonary embolism).

Objectively documented recurrent venous thromboembolism (either new or extended upper extremity deep vein thrombosis, proximal lower extremity deep vein thrombosis or pulmonary embolism) while taking systemic anticoagulation medication (Rivaroxaban).

Exclusion Criteria:

Previous hemorrhagic stroke Ischemic stroke in the last 3 months Severe renal impairment (CrCl rates < 30 ml/min) Active liver disease (any etiology) Concomitant use of any antiplatelet (aspirin, clopidogrel, prasugrel, ticagrelor, ticlopidine, etc.) Increased risk of bleeding (congenital or acquired) Uncontrolled SAH Gastrointestinal hemorrhage within the past year Anemia (Hb level < 10 g/dl) or thrombocytopenia (platelet count < 100 × 109/l) Pregnant or lactating women

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome The presence of thromboembolic events | 90 days
  Recurrent ipsilateral Deep vein thrombosis, Recurrent contralateral Deep vein thrombosis, Pulmonary emboli, Ischemic stroke and Myocardial infarction

SECONDARY OUTCOMES:
Major or clinically relevant nonmajor bleeding | 90 days
  The primary safety outcome was major or clinically relevant nonmajor bleeding according to the International Society on Thrombosis and Haemostasis (ISTH) criteria and Bleeding Academic Research Consortium (BARC)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano Del Seguro Social, Metepec, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No